CLINICAL TRIAL: NCT04151264
Title: Influence of the "Hypotension Probability Index" on the Number and Duration of Intraoperative and Postoperative Hypotension During Extended Surgical Procedures in ENT- and OM-Surgery
Brief Title: Influence of the "Hypotension Probability Index" on Intraoperative and Postoperative Hypotension in ENT- and OM-Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPI II
Record Dates: First submitted 2019-10-14; First posted 2019-11-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypotension; ENT Disease; Acute Kidney Injury; Anesthesia
Keywords: Hypotension; tumor of the oropharynx; tumor of the nasopharynx; creatinine
MeSH Terms: conditions — Hypotension; Otorhinolaryngologic Diseases; Acute Kidney Injury; Oropharyngeal Neoplasms; Nasopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized two arm study with two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): blinded HPI monitoring
- Intervention Arm (Active Comparator): HPI monitoring to predict hypotension
  Interventions: Device: Hypotension probability index (HPI)

INTERVENTIONS:
Device: Hypotension probability index (HPI) — The intervention group is managed with the HPI parameter to detect and possibly prevent hypotension during anaesthesia.
  Arms: Intervention Arm

SUMMARY:
The aim of the project is to investigate whether the use of the HPI can reduce the number and duration of intra- and postoperative hypotension in ventilated patients during and two hours after extensive surgery in the head and neck area compared to the established monitoring.

DETAILED DESCRIPTION:
Blood pressure monitoring displays a crucial part of anesthetic management. An intraoperative hypotension (IOH) is an unwanted complication that can occur during an anaesthetization or during the following duration of the surgery. Causes for this can be vasodilatation (e.g. due to medication), loss of blood volume (e.g. bleeding) or lack of inotropy (reduced left ventricular function, e.g. due to medication).

The main high-risk factors for intraoperative hypotension are age of the patient, pre-existing diseases (especially ASA 3 and higher), the duration of surgery, the urgency of the surgery (emergency surgery), antihypertensive long-term medication as well as combined anaesthesia (regional and general anaesthesia).

According to the examined collective, the definition of IOH and the level of training of the performing doctor we can monitor IOH in up to 100% of patients (depending on the data collection). Monk et al. show that the one-year mortality of patients undergoing surgery was elevated to 3.6% for every minute the systolic pressure was less than 80mmHg. Also, the risk of mortality was 1.4 higher if the MAP decreased <55mmHg. The consequence of IOH can be a critical reduction of the oxygen supply in the organs. Therefore, organs with low tolerance for hypoxia or a high necessity for oxygen are prone to hypotension induced complications. Those include ischemic stroke or myocardial ischemia (especially in patients with preexisting anemia), mostly happening to older or critical ill patients.

The extensive surgeries in ENT- and OM surgery are usually due to tumor diseases. The incidence for hypopharynx carcinoma is between 2-3/10.000 cases each year with an increasing tendency. The peak of this disease is in the 5.-6. decade of life. Causes for this are chronic noxae like alcohol and cigarettes. Numbers show, that the percentage of malignant tumors in the oral cavity and the pharynx in Germany in 2012 were at 3.7% with men and 1.6% with women in the entirety of incidence of malignant tumors. Especially these tumors require a radical resection also in the initial state of the disease which comes along with a long duration of surgery. The operative interventions include a radical resection of the tumor, neck dissection and if necessary a skin flap depending on the state of the tumor, TNM classification and status of lymph nodes. Complications that can occur with these types of surgery are (secondary) bleeding, stenosis, dyspnea, oedema of the mucosa, subcutaneous emphysema, dysphagia and aspiration. Because of the surgical treatment these patients require a postoperative sedation and ventilation. This enables the protection of the respiratory system when patients are at high risk for intra- or postoperative secondary bleeding and/or swelling. Also, the sedation will help not to imperil the success of the intervention (e.g. through coughing, pressure or choking).

The Hypotension Prediction Index (HPI) was developed by Edwards Lifesciences (Irvine, California, USA) and is certified in the US and Europe. As part of the Edwards Acumen Decision Support software suite, the HPI is based on the minimal invasive FloTrac IQ sensor. The HPI indicates the probability of an occurring hypotensive event. The software was developed using 20,000 cases of past patient events. If the upper limit of hypotension is reached, the software will alert the responsible physician.

The main outcome criteria are the numbers (n) and duration in minutes (t [min]) of intraoperative and postoperative hypotension. These are defined as MAP below 65 mmHg for more than one minute in ventilated patients with and without the use of HPI.

The secondary objective criteria are the following:

* Assumed reason for hypotension
* Amount of applied infusion volume (crystalloids, colloids, blood products and blood)
* Type and dose of applied vasopressors
* Type and dose of applied inotropic agents
* Acute Kidney Injury Risk Score

ELIGIBILITY:
Inclusion Criteria:

* extensive surgery in the head and neck area
* Age ≥ 18 years

Exclusion Criteria:

* Participation in another interventional study
* Pregnancy and nursing mothers
* Surgery without controlled ventilation
* Contraindication to invasive arterial pressure measurement
* Renal insufficiency KDIGO stage ≥ 3
* Congenital coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
number (n) of intraoperative and postoperative hypotension | until 4 hours after the end of surgery
  MAP below 65 mmHg for more than one minute in ventilated patients

SECONDARY OUTCOMES:
Applied volume in ml | until 4 hours after the end of surgery
  Amount of applied infusion volume (crystalloids, colloids, blood products and blood) in ml
Changes of catecholamine management | until 4 hours after the end of surgery
  Dosage of vasopressors and inotropes (in μg)
Duration of surgery | up to 24 hours
  cut-seam time
Fluid balance | until 4 hours after the end of surgery
  blood loss and urin output in ml
Hospital length of stay | up to 18 month
  Duration of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, Prof., Study Director — UKGM Giessen
Locations (1):
- University Clinic Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Bijker JB, Persoon S, Peelen LM, Moons KG, Kalkman CJ, Kappelle LJ, van Klei WA. Intraoperative hypotension and perioperative ischemic stroke after general surgery: a nested case-control study. Anesthesiology. 2012 Mar;116(3):658-64. doi: 10.1097/ALN.0b013e3182472320. PMID 22277949
- [Derived] Ali Akbari A, Koch C, Schmidt G, Schmermund D, Langer C, Edinger F, Denn SM, Markmann M, Sander M, Habicher M. Artificial intelligence-based predictive hemodynamic monitoring in conjunction with goal-directed therapy reduces duration, frequency, and severity of intraoperative hypotension in major maxillofacial and otolaryngological surgery-a prospective randomized controlled pilot trial. J Anesth Analg Crit Care. 2025 Dec 22;5(1):92. doi: 10.1186/s44158-025-00331-1. PMID 41423680
- See also: German Cancer Record — https://www.krebsdaten.de/Krebs/DE/Home/homepage_node.html
- See also: Edwards Information — https://www.edwards.com/de/devices/Hemodynamic-Monitoring/FloTrac